CLINICAL TRIAL: NCT01276080
Title: A Study to Evaluate A Study to Evaluate the Relative Bioavailability of Donepezil Hydrochloride 10 mg Tablets (OHM Laboratories, Inc., USA) Compared to ARICEPT® (Donepezil Hydrochloride)10 mg Tablets (Eisai Inc.) in Healthy Volunteers Under Non-Fasted Conditions
Brief Title: Bioequivalence Study of Donepezil Hydrochloride 10 mg Tablets Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Sponsor
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 10940308
Record Dates: First submitted 2011-01-11; First posted 2011-01-13 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-06

CONDITIONS: Healthy
MeSH Terms: interventions — Donepezil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Donepezil Hydrochloride 10 mg Tabletof OHM Laboratories, Inc.
  Interventions: Drug: Donepezil
- 2 (Active Comparator): ARICEPT® (donepezil hydrochloride) 10 mg Tablet of Eisai, Inc.
  Interventions: Drug: Donepezil

INTERVENTIONS:
Drug: Donepezil — 10 mg tablets

SUMMARY:
This open label, balanced, randomized, two-treatment, two-period, two-sequence, single dose crossover study was conducted to compare the relative bioavailability of equal doses of the test and reference products under non-fasted conditions.

DETAILED DESCRIPTION:
This open label, balanced, randomized, two-treatment, two-period, two-sequence, single dose crossover study was conducted to compare the relative bioavailability of equal doses of the test and reference products under non-fasted conditions. The study was conducted with 36 (31 completing) healthy adults in accordance with Protocol No. 10940308 (Revision 0). In each study period, a single 10 mg tablet of donepezil hydrochloride was administered to all subjects following a standardized high fat, high calorie breakfast, preceded by an overnight fast of at least 10 hours. The test formulation was donepezil hydrochloride 10 mg tablet (OHM Laboratories, Inc., USA a subsidiary of Ranbaxy Pharmaceuticals, Inc. USA) and the reference formulation was ARICEPT® (donepezil hydrochloride) 10 mg Tablets (Eisai Inc.). The subjects received the test product in one study period and the reference product in the other period; the order of administration was according to the dosing randomization schedule. Subjects were confined at the clinical facility from at least 10.5 hours prior to dosing until after the 24 hour blood collection. Subjects returned to the clinical facility for the 36, 48, and 72 hour blood sample collection. There was a 28-day interval between treatments.

Blood samples were collected pre-dose and at intervals over 72 hours after dosing in each period. The plasma samples from all subjects were shipped to Warnex Bioanalytical Services for determination of donepezil concentrations.

Statistical analysis was performed by Ranbaxy Laboratories Limited to compare the bioequivalence of the test formulation to the reference product. Bioequivalence was determined based on the confidence intervals for the major pharmacokinetic parameters, AUC0-72 and Cmax, for donepezil.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, 18 to 65 years of age (inclusive) and a Body Mass Index (BMI) 18 to 30 kg/m² inclusive. BMI will be calculated using Novum Pharmaceutical Research Services Standard Operating Procedures
2. Female subjects of child bearing potential must either abstain from sexual intercourse, or use a reliable non-hormonal method of contraception (e.g. condom with spermicide, IUD) for at least 30 days prior to dosing and during the duration of the study. The use of any type of hormonal contraception is not allowed.
3. Good health as determined by lack of clinically significant abnormalities in health assessments performed at screening.
4. Signed and dated informed consent form, which meets all criteria of current FDA regulations.

Exclusion Criteria:

1. Females who are pregnant, lactating or likely to become pregnant during the study
2. History of allergy or sensitivity to donepezil, other cholinesterase inhibitors, or history of any drug hypersensitivity or intolerance which, in the opinion of the Investigator, would compromise the safety of the subject or the study.
3. Significant history or current evidence of chronic infectious disease, system disorder or organ dysfunction.
4. Presence of gastrointestinal disease or history of malabsorption within the last year. Any history of gastrointestinal ulcers, bleeding or obstruction.
5. History of asthma or obstructive pulmonary disease.
6. History of psychiatric disorders occurring within the last two years that required hospitalization or medication.
7. Presence of a medical condition requiring regular treatment with prescription drugs (including hormonal contraceptives).
8. Use of pharmacologic agents known to significantly induce or inhibit drug-metabolizing enzymes within 30 days prior to dosing.
9. Receipt of any drug as part of a research study within 30 days prior to dosing.
10. Drug or alcohol addiction requiring treatment in the past 12 months.
11. Donation or significant loss of whole blood (480 ml or more) within 30 days or plasma within 14 days prior to dosing.
12. Positive test results for HIV, Hepatitis B surface antigen or Hepatitis C antibody.
13. Positive test results for drugs of abuse or alcohol at screening.
14. Positive serum pregnancy test.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-10; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Bioequivalence evaluation of Donepezil 10mg tablets | completed

CONTACTS AND LOCATIONS:
Locations (1):
- Novum Pharmaceutical Research Services, Las Vegas, Nevada, United States

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html